CLINICAL TRIAL: NCT06156904
Title: A Post-market Clinical Follow-up Investigation to Confirm the Performance and Safety of the Bone Substitute b.Bone in Extremities and Pelvis.
Brief Title: OSsIRIS Study - A Post-market Clinical Follow-up Investigation.
Acronym: OSsIRIS
Status: Recruiting | Type: Observational
Sponsor: GreenBone Ortho S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-GB002-22-0123
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Surgically Created Bone Defects or Bone Defects/Voids Resulting From Traumatic Injury
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bone grafting for the treatment of surgically created bone defects or bone defects/voids resulting from traumatic injury to promote healing in the pelvis, upper and lower extremities. — All patients enrolled in this clinical investigation will undergo a reconstruction of surgically created osseous defects or osseous defects resulting from traumatic injury to the bone as per the standard of care at the investigational sites. Patients will be treated with b.Bone which will be used as a bone substitute in isolation or as a graft expander to promote healing in the pelvis, upper and lower extremities.
  b.Bone is a bone substitute without initial mechanical properties, therefore it is to be used in conjunction with internal/external fixation devices suitable for primary stabilization.

SUMMARY:
This is a prospective, observational, non-randomized, multicenter, international post-market clinical follow-up investigation aiming to confirm the performance and safety of the bone substitute b.Bone after implantation in patients in isolation or as a graft expander requiring bone grafting for the treatment of surgically created bone defects or bone defects/voids resulting from traumatic injury to promote healing in the pelvis, upper and lower extremities. Patients enrolled in this clinical investigation will undergo orthopaedic surgery with b.Bone as recommended by the specialist and according to orthopaedic standard procedures. Patients will be evaluated preoperatively and at different time points after the surgery according to the standard practice of the sites. The expected schedule is at month 3, month 6 and month 12. Patients who require longer follow-up and could be subjected to metalwork removal will be evaluated up to 24 months. All safety data will be collected from patient inclusion to the end of the clinical investigation.

All study visits will coincide with any of the patient's routine clinical visits, without interfering with the investigator's clinical duties.

It is planned to enroll 135-193 patients from approximately 15 EU and UK sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is undergoing a standard of care bone grafting with b.Bone for the treatment of surgically created bone defects or bone defects resulting from traumatic injury in the extremities and pelvis according to the approved IFU.
2. Male or female patient ≥ 18 years old.
3. Patients willing and able to attend the standard of care follow-up visits and procedures.
4. Patients who have provided consent to participate in the clinical investigation and to the processing of personal data.

Exclusion Criteria:

1. Patients with any conditions in which b.Bone is not indicated according to the contraindications defined in the IFU of b.Bone
2. Patients who are currently enrolled in another clinical investigation/study that would directly interfere with the current clinical investigation, except when the patient is participating in a purely observational study with no associated treatments.
3. Woman who is pregnant or breast-feeding.
4. Patients who, in the opinion of the Investigator, have an existing condition that could affect their ability to complete patient reported questionnaires or be compliant with the standard of care follow-up visits and examinations for the duration of the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients both sexes requiring bone grafting with the synthetic bone substitute b.Bone, according to the standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Performance of b.Bone by determining the radiographic healing/union after surgery. | 12 months
  Number and rate of patients with successful bone healing/union observable by X-ray or CT scan.
  Radiologic images will be evaluated by the surgeon according to the modified radiographic Union Scale for Tibial fractures (mRUST) classification or the modified Neer classification when applicable.

SECONDARY OUTCOMES:
Clinical outcomes measured by patient-reported outcomes - Pain | Baseline and 3, 6 and 12 months
  Change in the patient-reported pain using the Visual Analoge Scale from baseline to month 3, month 6 and month 12 post-treatment.
  Patient-completed questionnaire scoring pain by using 10 cm line. Zero (0) indicates no pain at all and ten (10) the worst pain ever.
Clinical outcomes measured by patient-reported outcomes - Quality of Life | Baseline and 3, 6 and 12 months
  Change in the patient-reported Quality of Life assessed by Health Questionnaire from baseline to month 3, month 6 and month 12 post-treatment.
Evaluate the safety of b.Bone during the clinical investigation period - AE and SAE | Up to 24 months
  Number and rate of procedure and device-related adverse events (AEs) and Serious adverse events (SAEs) during the clinical investigation period.
Evaluate the safety of b.Bone during the clinical investigation period - rate of reinterventions | Up to 24 months
  Rate of reinterventions related to the treatment applied during the clinical investigation

OTHER OUTCOMES:
Exploratory outcomes: Evaluate the evolution over time of complementary radiographic parameter - bone formation | Up to 24 months
  Change of bone formation observable by X-ray/CT scan from the first evaluation immediately after b.Bone implantation through the observational period until the last available X-ray/CT scan.
Exploratory outcomes: Evaluate the evolution over time of complementary radiographic parameter - remodelling | Up to 24 months
  Change of remodelling observable by X-ray/CT scan from the first evaluation immediately after b.Bone implantation through the observational period until the last available X-ray/CT scan.
Exploratory outcomes: Evaluate the evolution over time of complementary radiographic parameter - material resorption | Up to 24 months
  Change of material resorption observable by X-ray/CT scan from the first evaluation immediately after b.Bone implantation through the observational period until the last available X-ray/CT scan.
Exploratory outcomes: Evaluate the performance of b.Bone on different anatomical sites of implantation. | Baseline and 3, 6 ,12, 24 months
  b.Bone performance on different subsets of patients depending on the anatomical site of implantation:
  * subset a: pelvis
  * subset b: upper extremities
  * subset c: lower extremities
  (The performance will be assessed as defined for the primary and secondary outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Alt, Dr, Principal Investigator — Director of the Trauma Surgery Department University Hospital Regensburg, Germany; Peter Giannoudis, Dr, Principal Investigator — Honorary Consultant Trauma & Orthopaedic Surgery, Leeds General Infirmary, United Kingdom
Locations (4):
- Germany (2):
  - BG Klinikum Unfallkrankenhaus Berlin, Berlin
  - Trauma Surgery Department - University Hospital Regensburg, Regensburg
- United Kingdom (2):
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Department of Trauma and Orthopaedic Surgery, Leeds General Infirmary, Leeds